CLINICAL TRIAL: NCT00633828
Title: Determinants for Peak Bone Mass, Skeletal Architecture, Fractures, Adipositas and Cardiovascular Risk Factors During Growth and Adulthood
Brief Title: Influence of External Factors on Skeletal Growth in Youth
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NKOISR10002
Record Dates: First submitted 2008-03-04; First posted 2008-03-12 (Estimated); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Fractures
Keywords: Bone Density; Bone mass; Bone mineral density; Bone structure; Cardiovascular risk factors; Fat Mass; Adiposity
MeSH Terms: conditions — Fractures, Bone; Obesity | interventions — Schools

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A Intervention group (Experimental): Increased physical education in primary school (daily)
  Interventions: Behavioral: Increased physical education in primary school (daily)
- B Control group (No Intervention): Normal physical education in primary school (typically once per week)

INTERVENTIONS:
Behavioral: Increased physical education in primary school (daily) — Increased physical education in primary school, 40 minutes per day
  Arms: A Intervention group

SUMMARY:
Objective:

Prospective study regulation in bone mass, size, architecture, cortical, trabecular bone, soft tissues and risk factors for cardiovascular disease at growth. Determine regulation by environmental factors. Evaluate how training affects the skeleton, soft tissues and cardiovascular risk factors during growth Material/Methods: (i) 500 children in one RCT´s with or without intervention with physical activity (daily scholl physical education) from school start to college. Annual evaluations

Importance:

The investigators provide increased understanding of the pathophysiology of osteoporosis by determine the mineralization, size- and architecture development during growth and adulthood. Evaluate if intervention program with exercise increase bone strength, muscle mass and reduce fatness and risk factor for cardiovascular disease.

Background:

Skeletal growth and the age related bone loss determine who will get osteoporosis (and fractures), but not only bone mass, also skeletal architecture and bone quality influence bone strength. Regulation of the traits differs where hormones, genetics and environmental factors continuously influence the development with different effect during different ages. It is thus imperative to determine the regulators of the traits and evaluate if these can be modified during growth.

Aim:

Study regulation of bone mass, size, architecture, cortical, trabecular, axial and appendicular bone and soft tissue during growth and aging; evaluate risk factors for cardiovascular disease; determine importance of environmental factors and hereditary factors.

Study Design/Method

Bunkeflo Cohort:

Prospective, controlled exercise intervention study annually following skeletal development in 500children from age 7.

Importance:

By evaluating skeletal mass/architecture separate we will increase the understanding of the pathophysiology of osteoporosis. The intervention study provide Evidence Based Information as regard the importance of physical activity during growth. The presented Strength Index, where we combine bone mass and skeletal architecture, may predict fractures better than only bone mass.

DETAILED DESCRIPTION:
Determinants for Peak Bone Mass, Skeletal Architecture, Fractures, Adipositas and Cardiovascular Risk Factors During Growth and Adulthood

Aim of the project:

In the THE BUNKEFLO COHORT we determine if the growing skeleton, fat mass and risk factors for cardiovascular disease irreversible can be influenced by environmental influences as exercise and disease.

Background:

Bone mass, cortical thickness and bone geometry independently contribute to bone strength, all regulated differently. Thus, the regulation must therefore be trait specific studied as to understand the pathophysiology of osteoporosis as osteoporosis may partly be the result of deficits occurring during growth. We must also better discriminate the different traits building the skeleton. Areal bone mineral density (aBMD), measured by dual X-ray absorptiometry (DXA) the clinically used estimation of bone mass, is an estimate only adjusted for the measured area, not the third dimension (the depth), but aBMD is often uncritically used as a measurement for the "true density". As to predict future fragility fracture, aBMD is acceptable, but for the understanding of reduced bone strength, we must separate the estimation into bone mass, the amount of bone within the skeletal envelope, bone size and skeletal structure (architecture) as these traits are independent associated with fractures.

Preliminary results from our group:

Bone loss by ageing is partly compensated by increased bone size, partly preserving bone strength. This is of relevance as a Strength Index, taking both bone size and bone mass into account, probably predict future fractures better than bone mass. Two years daily school gymnastics enhanced bone mass and bone size, reduce the fatness and cardiovascular risk factors for disease. Exercise increase bone mass also after puberty but the benefit is lost with cessation of exercise. In spite of this have elderly former active individuals less fractures than inactive people.

Research Questions Following Our Hypothesis:

1. Will separate evaluation of skeletal growth in bone mineral acquisition and skeletal architecture identify different pathogenetic risk cohorts for fracture?
2. Could an exercise intervention program within a school affect the skeletal growth, fat content soft and muscle strength in growing children and reduce risk for cardiovascular disease? (BUNKEFLO STUDY)?

Methods: Skeletal Evaluation: Dual X-ray absorptiometry (DXA, Lunar DPX-L and Lunar Pixi): Quantitative bone mass (aBMD) total body, femoral neck, lumbar spine and regional. Special software determines cortical width, medullar width, cortical density and trabecular density in mid femur. vBMD and skeletal size can be evaluated from existing measurement in femoral neck and third lumbar vertebrae from DXA scan by the method described by Carter. Ultrasound (Lunar Achilles): Qualitative bone mass (aBMD) and bone width calcaneus. Peripheral computed tomography (pQCT): Bone mass, bone size and skeletal structure. Finite element analyses: skeletal strength. Digital radiographs of the hand: Bone size and cortical thickness. Soft tissue Evaluation: DXA (Lunar DPX-L): Quantitative lean body mass and fat mass. Peripheral computed tomography (pQCT): Quantitative lean body mass and fat mass. Muscle function: Cybex apparatus: Qualitative muscle strength in lower extremities. Balance plate and physiotherapists test: Qualitative muscle capacity. Anthropometric evaluation: Electronic scale: Body weight. Holstein Stadiometer: Sitting and standing height. Harpender stadiometer: Segmental extremity length and width. Pubertal status: Tanner. Environmental Evaluation: Questionnaire: life-style, exercise history, nutrition, and hereditary factors. Bone metabolism: Bone formation: Alkaline phosphatase (ALP), isoenzyme of bone specific ALP, osteocalcin (bone GLA protein), procollagen 1 C-terminal propeptic (P1CP). Bone resorption: Hydroxyproline, pyridinoline, deoxypyridinoline, carboxytelopeptid region (ICTP) and aminotelopeptid region (NTX) in blood and urine. Genetics: Polymorphism of Vitamin D receptor gene (VDR), oestrogen receptor gene (ER), androgen receptor gene (AR), human growth hormone gene (GH 1), collagen 1 A gene (COLL1A) and additional bone related genes that will occur the next years. Hormones: Growth hormone, IGF-1, testosterone, estradiol, luteinisating hormone, follicle stimulating hormone, sex hormone binding globulin (SHBG), androstenedione, dehydroepiandrostenedione (DHEAS). Fractures: The fractures are registered in the files at the Dept. of Radiology, MAS where referrals, reports and films are saved since last century. Questionnaire: Epidemiologic fracture screening. Physiologic Evaluation: Blood pressure (rest): Upper right arm. Bicycle test: Max working capacity by evaluating VO2 MAX. and CO2 production in breath. Bio impedance: Fat percent in total body. Spirometry: Static and dynamic lung function measured by the IOS-method. Ultrasound: Volume and wall thickness of heart. Accelerometer: Number of steps during four days is measured within this minicomputer fastened at the wrist belt (evaluate the objective activity level). Blood Evaluation: Lipid profile and glucose - risk factors for cardiovascular disease and metabolic syndrome.

Probands - Work plan:

A. Determinants of Peak Bone Mass/Size/Architecture, Soft Tissue Development and Risk Factors for Cardiovascular disease During Growth Question: Regulation affecting growth and peak bone mass? Can increased exercise increase bone mass, reduce fatness and risk factors for cardiovascular disease? Could individuals with high risk for fractures be predicted already in early ages? Hypothesis: Changes in environmental factors can increase peak bone mass, reduce fatness and risk factors for future cardiovascular disease. Bone mass "track" so that we could already in young years identify individuals with high risk for fractures.

Study cohorts: a. THE BUNKEFLO STUDY: N=500, aged 7, 8, 9, 12 and 15 years at baseline. In the RCT part of the study: n=310 aged 7-8 at baseline. Half with physical activity and health education as intervention, half controls, all annually followed during primary school. Several other scientific institutions from the University of Lund participate as Department of Physiotherapy, Clinical Physiology, Nutritional, Paediatrics, Child Psychiatry, Teacher Training College, and Dental School, all with separate projects within the RCT. Time plan: Baseline measurements in 1999-2000, with annual follow-up measurements throughout the Swedish nine-year primary school. After that, one follow-up during the last year of secondary school (12th grade), and one follow-up at age 23-25.

Relevance:

The studies will increase the understanding of the pathophysiology of osteoporosis. The Strength Index should possibly replace a bone mass measurement in the fracture risk assessment. The intervention studies will provide Evidence Based Information for the importance of exercise.

ELIGIBILITY:
Inclusion Criteria:

* All included within the classes, population based cohort

Exclusion Criteria:

* None

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 500 (Actual)
Dates: Start 1999-08 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2050-12-31 (Estimated)

PRIMARY OUTCOMES:
BMD total body, femoral neck and lumbar spine (L2-L4) measured by Dual Energy X Ray Absorbtiometry | 15 years

SECONDARY OUTCOMES:
Bone mineral content (BMC) measured by DEXA and PQCT | 15 years
Bone mineral density (aBMD) measured by DEXA, ultrasound and PQCT | 15 years
Volumetric bone density (vBMD) measured by DEXA and PQCT | 15 years
Trabecular BMD measured by PQCT | 15 years
Cortical BMD measured by PQCT | 15 years
Periosteal diameter measured by DEXA andPQCT | 15 years
Medullary diameter measured by PQCT | 15 years
Cross sectional area (CSA) measured by PQCT | 15 years
Hip strength analysis (HSA) measured by DEXA | 15 years
Speed of sound (SOS) measured by quantitative ultrasound | 15 years
Broadband attenuation (BUA) measured by quantitative ultrasound | 15 years
Isodynamic muscle strength in thigh (knee extension and knee flexion, functional results of physiotherapy tests and CYBEX apparatus | 15 years
Fracture incidence determined through the radiographica archives in Malmö | 15 years
DXA derived fat content and lean body mass from total body scan | 15 years
Cardiovascular risk factors | 15 years
  Risk factors measured as
  * patients movement over 4 days measured by Accelerometer
  * blood pressure
  * heart volume by ultrasound
  * lung function monitored by spirometer
  * max VO2 from bicycle test

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Karlsson, M.D., Ph.D., Principal Investigator — Clinical and Molecular Osteoporosis Research Unit, Department of Clinical Sciences and Orthopaedic Surgery Lund University, Skåne Universíty Hospital

REFERENCES:
- [Derived] Rosengren BE, Lindgren E, Jehpsson L, Dencker M, Karlsson MK. Musculoskeletal Benefits from a Physical Activity Program in Primary School are Retained 4 Years after the Program is Terminated. Calcif Tissue Int. 2021 Oct;109(4):405-414. doi: 10.1007/s00223-021-00853-0. Epub 2021 Apr 29. PMID 33914096
- [Derived] Lahti A, Rosengren BE, Dencker M, Nilsson JA, Karlsson MK. Socioecological and biological associations of lower levels of physical activity in 8-year-old children: a 2-year prospective study. BMJ Open Sport Exerc Med. 2019 Nov 21;5(1):e000597. doi: 10.1136/bmjsem-2019-000597. eCollection 2019. PMID 31803494
- [Derived] Stenevi Lundgren S, Rosengren BE, Dencker M, Nilsson JA, Karlsson C, Karlsson MK. Low physical activity is related to clustering of risk factors for fracture-a 2-year prospective study in children. Osteoporos Int. 2017 Dec;28(12):3373-3378. doi: 10.1007/s00198-017-4203-0. Epub 2017 Sep 15. PMID 28913570
- [Derived] Coster ME, Fritz J, Nilsson JA, Karlsson C, Rosengren BE, Dencker M, Karlsson MK. How does a physical activity programme in elementary school affect fracture risk? A prospective controlled intervention study in Malmo, Sweden. BMJ Open. 2017 Feb 23;7(2):e012513. doi: 10.1136/bmjopen-2016-012513. PMID 28235964
- [Derived] Detter F, Nilsson JA, Karlsson C, Dencker M, Rosengren BE, Karlsson MK. A 3-year school-based exercise intervention improves muscle strength - a prospective controlled population-based study in 223 children. BMC Musculoskelet Disord. 2014 Oct 27;15:353. doi: 10.1186/1471-2474-15-353. PMID 25345446
- [Derived] Lofgren B, Dencker M, Nilsson JA, Karlsson MK. A 4-year exercise program in children increases bone mass without increasing fracture risk. Pediatrics. 2012 Jun;129(6):e1468-76. doi: 10.1542/peds.2011-2274. Epub 2012 May 28. PMID 22641757